CLINICAL TRIAL: NCT03216733
Title: Randomized Clinical Comparison of a Combined Sirolimus Eluting and Endothelial Progenitor Cell COMBO Stent With a Sirolimus-eluting OSIRO Stent in Patients Treated With Percutaneous Coronary Intervention - The SORT-OUT X Study
Brief Title: SORT OUT X - Combo Stent Versus ORSIRO Stent
Acronym: SORT OUT X
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Biotronik SE & Co. KG (Industry); OrbusNeich (Industry)
Responsible Party: Principal Investigator, Lars Jakobsen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-38-17
Record Dates: First submitted 2017-07-04; First posted 2017-07-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Coronary Heart Disease; Angina Pectoris; Myocardial Infarction
Keywords: DES; Angina pectoris; Stent
MeSH Terms: conditions — Coronary Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMBO (Experimental): PCI with COMBO stent
  Interventions: Device: COMBO
- ORSIRO (Active Comparator): PCI with ORSIRO stent
  Interventions: Device: ORSIRO

INTERVENTIONS:
Device: COMBO — PCI with COMBO stent
  Other Names: Combined Sirolimus eluting and endothelial progenitor cell stent
  Arms: COMBO
Device: ORSIRO — PCI with ORSIRO stent
  Other Names: Sirolimus-eluting stent
  Arms: ORSIRO

SUMMARY:
The aim of the Danish Organisation for randomised trials with clinical outcome (SORT OUT) is to compare the safety and efficacy of the ComboTM stent and Orsiro™ stent in the treatment of unselected patients with ischemic heart disease, using registry detection of clinically driven events.

DETAILED DESCRIPTION:
Randomized Clinical Comparison of a Combined Sirolimus Eluting and endothelial progenitor cell COMBO Stent with a Sirolimus-eluting OSIRO stent in Patients Treated with Percutaneous Coronary Intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years who are eligible for treatment with one or several drug-eluting coronary stents at Rigshospitalet or one of the three heart centers in Aarhus, Odense and Aalborg can be included in the study.
* The patients will be treated in accordance with the criteria applicable at the individual sites.
* The investigators plan to include 3,140 patients.

Exclusion Criteria:

* Age < 18 years
* The patient does not wish to participate
* The patient is not able to consent to randomization (eg intubated patients)
* The patient do not speak Danish
* The patient is already included in this study
* The patient is already participating in other stent studies
* Life expectancy <1 year
* Allergic to aspirin, clopidogrel, prasugrel or ticagrelor
* Allergic to sirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3148 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-related Target Lesion Failure (TLF) The composite of cardiac death, target-vessel myocardial infarction (MI), or ischemia-driven target-lesion revascularization | Within 12 months
  Analysing the Kaplan-Meier method. Hazard ratios between groups will be calculated using a Cox proportional hazard model and the primary endpoint in the two per protocol treated groups will be compared with an upper one-sided 95% confidence interval.
  Patients treated with the OsiroTM stent will be used as the reference group
Target Lesion Revascularisation (TLR) | Within 12 months
  Repeat/new revascularization (PCI or CABG) within the stent or within a 5-mm border proximal or distal to the stent. (Angina, CCS > 1 related to the index lesion/vessel and diameter stenosis ≥ 50%. Diameter stenosis will be assessed by eyeballing, FFR <0.80, or iFR< 0.90). TLR will be clinically driven.

SECONDARY OUTCOMES:
Individual components of the primary end point comprise the secondary end points | Clinical follow-up will be continued through 5 years
  cardiac death; MI; clinically indicated TLR; all death (cardiac and noncardiac) and target vessel revascularisation (TVR); definite, probable, possible, and overall stent thrombosis according to the Academic Research Consortium definition (22); and a patient-related composite end point (all death, all MI (including procedure related MI), or any revascularization). For continuous variables, the difference between the treatment groups will be evaluated using Wilcoxon's rank-sum test. For discrete variables, the differences will be given as numbers and in percentages and will be analyzed using Fisher's exact test. Two-sided test will be used, and a pvalue of 0.05 considered significant.
Cardiac death | Through 5 years
MI | Through 5 years
  The acute MI diagnosis follows "The Joint ESC/ACCF/AHA/WHF Task Force on "Third Universal Definition of MI" (23), which has been adapted by Academy Research Consortium (22).
  In cases of updates of the definition of MI, the latest definition will be used.
Clinically indicated TLR | Through 5 years
  Angina, CCS > 1 related to the index lesion/vessel and diameter stenosis ≥ 50%. Diameter stenosis will be assessed by eyeballing, FFR <0.80, or iFR< 0.90.
All death | Through 5 years
  Cardiac and noncardiac
TVR | Through 5 years
  Angina, CCS > 1 related to the index lesion/vessel and diameter stenosis ≥ 50%. Diameter stenosis will be assessed by eyeballing, FFR <0.80, or iFR< 0.90.
Stent thrombosis | Through 5 years
  Definite, probable, possible and overall according to the Academic Research Consortium definition (22)
Patient-related composite end point | Through 5 years
  All death, all MI (including procedure related MI) or any revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jakobsen, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Department of Cardiology, Aalborg
  - Aarhus University Hospital, Skejby, Aarhus N
  - Rigshospitalet, Hjertecentret, Copenhagen
  - Odense Unversity Hospital, Department of Cardiology, Odense C

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakobsen L, Christiansen EH, Freeman P, Kahlert J, Veien K, Maeng M, Raungaard B, Ellert J, Villadsen AB, Kristensen SD, Christensen MK, Terkelsen CJ, Aaroe J, Thim T, Lassen JF, Hougaard M, Eftekhari A, Jensen RV, Stottrup NB, Rasmussen JG, Junker A, Jensen SE, Hansen HS, Jensen LO. Dual-therapy CD34 antibody-covered sirolimus-eluting COMBO stents versus sirolimus-eluting Orsiro stents in patients treated with percutaneous coronary intervention: the three-year outcomes of the SORT OUT X randomised clinical trial. EuroIntervention. 2023 Oct 23;19(8):676-683. doi: 10.4244/EIJ-D-23-00330. PMID 37584207
- [Derived] Jakobsen L, Christiansen EH, Freeman P, Kahlert J, Veien K, Maeng M, Raungaard B, Ellert J, Villadsen AB, Kristensen SD, Ahlehoff O, Christensen MK, Terkelsen CJ, Erik Botker H, Aaroe J, Thim T, Thuesen L, Aziz A, Eftekhari A, Jensen RV, Stottrup NB, Rasmussen JG, Junker A, Jensen SE, Hansen HS, Jensen LO. Randomized Clinical Comparison of the Dual-Therapy CD34 Antibody-Covered Sirolimus-Eluting Combo Stent With the Sirolimus-Eluting Orsiro Stent in Patients Treated With Percutaneous Coronary Intervention: The SORT OUT X Trial. Circulation. 2021 Jun;143(22):2155-2165. doi: 10.1161/CIRCULATIONAHA.120.052766. Epub 2021 Apr 7. PMID 33823606
- [Derived] Jakobsen L, Christiansen EH, Maeng M, Kristensen SD, Botker HE, Terkelsen CJ, Madsen M, Raungaard B, Jensen SE, Christensen MK, Hansen HS, Jensen LO. Randomized clinical comparison of the dual-therapy CD34 antibody-covered sirolimus-eluting Combo stent with the sirolimus-eluting Orsiro stent in patients treated with percutaneous coronary intervention: Rationale and study design of the Scandinavian Organization for Randomized Trials with Clinical Outcome (SORT OUT) X trial. Am Heart J. 2018 Aug;202:49-53. doi: 10.1016/j.ahj.2018.04.019. Epub 2018 May 5. PMID 29807307